CLINICAL TRIAL: NCT05034835
Title: Impact of Compression Garments on Neuropathic-looking Pain in Patients With Complex Regional Pain Syndrome (CRPS) of the Upper Limbs.
Brief Title: Impact of Compression Garments on Pain in Patients With Complex Regional Pain Syndrome of the Upper Limbs.
Acronym: VECODON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Mutualiste de Rééducation et de Réadaptation Fonctionnelles de Kerpape (Other)
Collaborators: Clinique Mutualiste Lorient (Unknown); Fondation Rothschild Paris (Other); Groupement des Hôpitaux de l'Institut Catholique de Lille (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-A00657-32
Record Dates: First submitted 2021-08-26; First posted 2021-09-05 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Complex Regional Pain Syndromes
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Intervention Model Description: This research is part of a Research Involving the Human Person of the interventional type (RIPH1) and relates to a class I medical device (MD).
  This is a single-center, controlled, randomized, open-label, superiority study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- With compression garments (Experimental): Usual care in day hospitals, i.e. 3 occupational therapy sessions / week for 3 months, with the usual protocol of desensitization by Aquaroll (hydro-massage ball device) and by Vibralgic (device generating electronic transcutaneous vibrations) + wearing a compression garment for 3 months.
  Interventions: Device: usual treatment with compression garments (CERECARE)
- Without compression garments (Other): Usual care in day hospitals, i.e. 3 occupational therapy sessions / week for 3 months, with the usual protocol of desensitization by Aquaroll (hydro-massage ball device) and by Vibralgic (device generating electronic transcutaneous vibrations).
  Interventions: Other: usual treatment without compression garments (CERECARE)

INTERVENTIONS:
Device: usual treatment with compression garments (CERECARE) — For 3 months, the pain will be assessed every week, tolerance and compliance with compression garments will also be monitored. Participants will be reviewed specifically at a follow-up consultation for the 6-month and 1-year study. Various assessments will be carried out during these visits : assessment of pain, range of motion, muscle strength, sensitivity test, assessment of anxiety, depression and even quality of life.
  Arms: With compression garments
Other: usual treatment without compression garments (CERECARE) — For 3 months, the pain will be assessed every week, tolerance and compliance with compression garments will also be monitored. Participants will be reviewed specifically at a follow-up consultation for the 6-month and 1-year study. Various assessments will be carried out during these visits : assessment of pain, range of motion, muscle strength, sensitivity test, assessment of anxiety, depression and even quality of life.
  Arms: Without compression garments

SUMMARY:
The aim is to study another alternative for the treatment of pain in people with CRPS. Indeed, the TRAB / Medullary occupational therapy department of the CMRRF in Kerpape used compression garments to reduce edema when it was present.In the case of CRPS of the upper limbs, gloves or compression sleeves are used to decrease the edema which is sometimes associated, although they are not supported for this indication. In this context, our clinical experience leads us to believe that there would also be some efficacy in neuropathic pain, this improvement being regularly described by patients.This study is expected to show a notable reduction in neuropathic pain thanks to the wearing of a compression garment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CRPS of the upper limb with neuropathic pain

  * Diagnosis of CRPS according to the Budapest criteria
  * Diagnosis of neuropathic pain according to DN4
* CRPS evolving for more than 3 months
* No phlebitis or open sores on the upper limbs
* Patient consent to participate in the study
* No modification of his drug treatment for 1 month
* Affiliation to a social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* Patient under guardianship, curatorship or safeguard of justice
* Psychiatric pathology altering the ability to consent
* Severe cognitive disorders that do not allow the patient to assess his pain
* Skin pathology preventing the wearing of the compression garment
* Patient who has previously worn a compression garment
* History of vascular disorders of the upper limbs, lymph node dissection, or any other pathology that can lead to edema regardless of CRPS
* Known allergy to one of the components of the compression garments of the Cerecare brand
* Declared pregnancy, breastfeeding woman or woman of childbearing potential without contraception
* Inability to put on the compression garment alone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
The evolution of pain through Visual Analog Scale (VAS), measured every week for 3 months in the last 24 hours and in the last 7 days | up to 3 months
  The VAS is a self-rated scale. It comes in the form of a 10 cm plastic ruler graduated in mm. On the face presented to the patient is a cursor which he moves along a straight line, one end of which corresponds to "No pain" and the other to "Maximum pain imaginable". The patient should, along this line, position the cursor where the pain is best located. On the other side, there are millimeter graduations seen only by the caregiver. The position of the cursor mobilized by the patient makes it possible to read the intensity of the pain, which is measured in mm.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | At 6 months
  The VAS is a self-rated scale. It comes in the form of a 10 cm plastic ruler graduated in mm. On the face presented to the patient is a cursor which he moves along a straight line, one end of which corresponds to "No pain" and the other to "Maximum pain imaginable". The patient should, along this line, position the cursor where the pain is best located. On the other side, there are millimeter graduations seen only by the caregiver. The position of the cursor mobilized by the patient makes it possible to read the intensity of the pain, which is measured in mm.
Visual Analog Scale (VAS) | At 1 year
  The VAS is a self-rated scale. It comes in the form of a 10 cm plastic ruler graduated in mm. On the face presented to the patient is a cursor which he moves along a straight line, one end of which corresponds to "No pain" and the other to "Maximum pain imaginable". The patient should, along this line, position the cursor where the pain is best located. On the other side, there are millimeter graduations seen only by the caregiver. The position of the cursor mobilized by the patient makes it possible to read the intensity of the pain, which is measured in mm.
Neuropathic Pain Symptom Inventory (NPSI) | Day 0
  It's a tool developed and validated in French, composed of 12 items. It provides an overall score and 5 sub-scores
Neuropathic Pain Symptom Inventory (NPSI) | At 1,5 months
  It's a tool developed and validated in French, composed of 12 items. It provides an overall score and 5 sub-scores
Neuropathic Pain Symptom Inventory (NPSI) | At 3 months
  It's a tool developed and validated in French, composed of 12 items. It provides an overall score and 5 sub-scores
Neuropathic Pain Symptom Inventory (NPSI) | At 6 months
  It's a tool developed and validated in French, composed of 12 items. It provides an overall score and 5 sub-scores
Neuropathic Pain Symptom Inventory (NPSI) | At 1 year
  It's a tool developed and validated in French, composed of 12 items. It provides an overall score and 5 sub-scores
Modification of analgesic drug treatment | Day 0
  The increase or decrease in doses between each visit will be collected by the doctor. He can rely on the booklet filled out by the patient.
Modification of analgesic drug treatment | At 1,5 months
  The increase or decrease in doses between each visit will be collected by the doctor. He can rely on the booklet filled out by the patient.
Modification of analgesic drug treatment | At 3 months
  The increase or decrease in doses between each visit will be collected by the doctor. He can rely on the booklet filled out by the patient.
Modification of analgesic drug treatment | At 6 months
  The increase or decrease in doses between each visit will be collected by the doctor. He can rely on the booklet filled out by the patient.
Modification of analgesic drug treatment | At 1 year
  The increase or decrease in doses between each visit will be collected by the doctor. He can rely on the booklet filled out by the patient.
Measurement of range of motion | Day 0
  The range of motion is measured exploratory at different levels, for both sides:
  * Wrist range of motion, measured using posture foam and goniometer. This measures the amplitude in flexion, extension, radial tilt, ulnar tilt, and pronation and supination, both passively and actively.
  * Pulp-palm and pulp palmar fold distances of the fingers, measured using wedges of different lengths. One measurement is made per finger
  * Kapandji score, which is a score out of 10 based on achievable opposition for the thumb. 0 being the lowest score and 10 a normal score.
Measurement of range of motion | At 1,5 months
  The range of motion is measured exploratory at different levels, for both sides:
  * Wrist range of motion, measured using posture foam and goniometer. This measures the amplitude in flexion, extension, radial tilt, ulnar tilt, and pronation and supination, both passively and actively.
  * Pulp-palm and pulp palmar fold distances of the fingers, measured using wedges of different lengths. One measurement is made per finger
  * Kapandji score, which is a score out of 10 based on achievable opposition for the thumb. 0 being the lowest score and 10 a normal score.
Measurement of range of motion | At 3 months
  The range of motion is measured exploratory at different levels, for both sides:
  * Wrist range of motion, measured using posture foam and goniometer. This measures the amplitude in flexion, extension, radial tilt, ulnar tilt, and pronation and supination, both passively and actively.
  * Pulp-palm and pulp palmar fold distances of the fingers, measured using wedges of different lengths. One measurement is made per finger
  * Kapandji score, which is a score out of 10 based on achievable opposition for the thumb. 0 being the lowest score and 10 a normal score.
Measurement of range of motion | At 6 months
  The range of motion is measured exploratory at different levels, for both sides:
  * Wrist range of motion, measured using posture foam and goniometer. This measures the amplitude in flexion, extension, radial tilt, ulnar tilt, and pronation and supination, both passively and actively.
  * Pulp-palm and pulp palmar fold distances of the fingers, measured using wedges of different lengths. One measurement is made per finger
  * Kapandji score, which is a score out of 10 based on achievable opposition for the thumb. 0 being the lowest score and 10 a normal score.
Measurement of range of motion | At 1 year
  The range of motion is measured exploratory at different levels, for both sides:
  * Wrist range of motion, measured using posture foam and goniometer. This measures the amplitude in flexion, extension, radial tilt, ulnar tilt, and pronation and supination, both passively and actively.
  * Pulp-palm and pulp palmar fold distances of the fingers, measured using wedges of different lengths. One measurement is made per finger
  * Kapandji score, which is a score out of 10 based on achievable opposition for the thumb. 0 being the lowest score and 10 a normal score.
Measurement of muscle strength in both hands | Day 0
  * the JAMAR® hydraulic hand dynamometer: measurement of the gripping force in kilograms
  * the PINCH® hydraulic pinch gauge: measures the pinch force in kilograms
Measurement of muscle strength in both hands | At 1,5 months
  * the JAMAR® hydraulic hand dynamometer: measurement of the gripping force in kilograms
  * the PINCH® hydraulic pinch gauge: measures the pinch force in kilograms
Measurement of muscle strength in both hands | At 3 months
  * the JAMAR® hydraulic hand dynamometer: measurement of the gripping force in kilograms
  * the PINCH® hydraulic pinch gauge: measures the pinch force in kilograms
Measurement of muscle strength in both hands | At 6 months
  * the JAMAR® hydraulic hand dynamometer: measurement of the gripping force in kilograms
  * the PINCH® hydraulic pinch gauge: measures the pinch force in kilograms
Measurement of muscle strength in both hands | At 1 year
  * the JAMAR® hydraulic hand dynamometer: measurement of the gripping force in kilograms
  * the PINCH® hydraulic pinch gauge: measures the pinch force in kilograms
Measurement of hand circumference | Day 0
  The circumference of the hand is measured in different places. A total of 15 measurements are taken. Both hands are measured.
  The analysis will be based on the difference of the sum of the 15 measures for each of the hands.
Measurement of hand circumference | At 1,5 months
  The circumference of the hand is measured in different places. A total of 15 measurements are taken. Both hands are measured.
  The analysis will be based on the difference of the sum of the 15 measures for each of the hands.
Measurement of hand circumference | At 3 months
  The circumference of the hand is measured in different places. A total of 15 measurements are taken. Both hands are measured.
  The analysis will be based on the difference of the sum of the 15 measures for each of the hands.
Measurement of hand circumference | At 6 months
  The circumference of the hand is measured in different places. A total of 15 measurements are taken. Both hands are measured.
  The analysis will be based on the difference of the sum of the 15 measures for each of the hands.
Measurement of hand circumference | At 1 year
  The circumference of the hand is measured in different places. A total of 15 measurements are taken. Both hands are measured.
  The analysis will be based on the difference of the sum of the 15 measures for each of the hands.
Saint-Antoine Pain Questionnaire (QDSA) | Day 0
  Illustrating the different components of pain, the QDSA (French version of the Mac Gill Pain Questionnary-MPQ) essentially allows a qualitative assessment of chronic pain, in particular neuropathic pain. It is a questionnaire of 58 qualifying words divided into subclasses: sensory pain on the one hand, affective and emotional pain on the other. The patient is asked to select the adjectives corresponding to his pain and then to note them from 0 (absent) to 4 (very strong). This self-assessment scale makes it possible in clinical practice to specify the involvement of the sensory and the emotional in pain intensity.
Saint-Antoine Pain Questionnaire (QDSA) | At 1,5 months
  Illustrating the different components of pain, the QDSA (French version of the Mac Gill Pain Questionnary-MPQ) essentially allows a qualitative assessment of chronic pain, in particular neuropathic pain. It is a questionnaire of 58 qualifying words divided into subclasses: sensory pain on the one hand, affective and emotional pain on the other. The patient is asked to select the adjectives corresponding to his pain and then to note them from 0 (absent) to 4 (very strong). This self-assessment scale makes it possible in clinical practice to specify the involvement of the sensory and the emotional in pain intensity.
Saint-Antoine Pain Questionnaire (QDSA) | At 3 months
  Illustrating the different components of pain, the QDSA (French version of the Mac Gill Pain Questionnary-MPQ) essentially allows a qualitative assessment of chronic pain, in particular neuropathic pain. It is a questionnaire of 58 qualifying words divided into subclasses: sensory pain on the one hand, affective and emotional pain on the other. The patient is asked to select the adjectives corresponding to his pain and then to note them from 0 (absent) to 4 (very strong). This self-assessment scale makes it possible in clinical practice to specify the involvement of the sensory and the emotional in pain intensity.
Saint-Antoine Pain Questionnaire (QDSA) | At 6 months
  Illustrating the different components of pain, the QDSA (French version of the Mac Gill Pain Questionnary-MPQ) essentially allows a qualitative assessment of chronic pain, in particular neuropathic pain. It is a questionnaire of 58 qualifying words divided into subclasses: sensory pain on the one hand, affective and emotional pain on the other. The patient is asked to select the adjectives corresponding to his pain and then to note them from 0 (absent) to 4 (very strong). This self-assessment scale makes it possible in clinical practice to specify the involvement of the sensory and the emotional in pain intensity.
Saint-Antoine Pain Questionnaire (QDSA) | At 1 year
  Illustrating the different components of pain, the QDSA (French version of the Mac Gill Pain Questionnary-MPQ) essentially allows a qualitative assessment of chronic pain, in particular neuropathic pain. It is a questionnaire of 58 qualifying words divided into subclasses: sensory pain on the one hand, affective and emotional pain on the other. The patient is asked to select the adjectives corresponding to his pain and then to note them from 0 (absent) to 4 (very strong). This self-assessment scale makes it possible in clinical practice to specify the involvement of the sensory and the emotional in pain intensity.
Cartographic assessment of pain | Day 0
  The cartographic assessment of pain is carried out following the QDSA. Using schematic representations of the hand (dorsal face and palmar face for each hand), the patient locates and describes his pain.
Cartographic assessment of pain | At 1,5 months
  The cartographic assessment of pain is carried out following the QDSA. Using schematic representations of the hand (dorsal face and palmar face for each hand), the patient locates and describes his pain.
Cartographic assessment of pain | At 3 months
  The cartographic assessment of pain is carried out following the QDSA. Using schematic representations of the hand (dorsal face and palmar face for each hand), the patient locates and describes his pain.
Cartographic assessment of pain | At 6 months
  The cartographic assessment of pain is carried out following the QDSA. Using schematic representations of the hand (dorsal face and palmar face for each hand), the patient locates and describes his pain.
Cartographic assessment of pain | At 1 year
  The cartographic assessment of pain is carried out following the QDSA. Using schematic representations of the hand (dorsal face and palmar face for each hand), the patient locates and describes his pain.
Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire | Day 0
  This is a subjective self-assessment questionnaire of the overall functional capacity of the two upper limbs, composed of 30 items, rated from 1 to 5 depending on the difficulty of the task described, leading to a score out of 100.
Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire | At 1,5 months
  This is a subjective self-assessment questionnaire of the overall functional capacity of the two upper limbs, composed of 30 items, rated from 1 to 5 depending on the difficulty of the task described, leading to a score out of 100.
Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire | At 3 months
  This is a subjective self-assessment questionnaire of the overall functional capacity of the two upper limbs, composed of 30 items, rated from 1 to 5 depending on the difficulty of the task described, leading to a score out of 100.
Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire | At 6 months
  This is a subjective self-assessment questionnaire of the overall functional capacity of the two upper limbs, composed of 30 items, rated from 1 to 5 depending on the difficulty of the task described, leading to a score out of 100.
Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire | At 1 year
  This is a subjective self-assessment questionnaire of the overall functional capacity of the two upper limbs, composed of 30 items, rated from 1 to 5 depending on the difficulty of the task described, leading to a score out of 100.
Hospital Anxiety and Depression (HAD) Scale | Day 0
  It comprises 14 items, allowing the obtaining of 2 scores out of 21 points, corresponding to the dimensions of anxiety and depression
Hospital Anxiety and Depression (HAD) Scale | At 1,5 months
  It comprises 14 items, allowing the obtaining of 2 scores out of 21 points, corresponding to the dimensions of anxiety and depression
Hospital Anxiety and Depression (HAD) Scale | At 3 months
  It comprises 14 items, allowing the obtaining of 2 scores out of 21 points, corresponding to the dimensions of anxiety and depression
Hospital Anxiety and Depression (HAD) Scale | At 6 months
  It comprises 14 items, allowing the obtaining of 2 scores out of 21 points, corresponding to the dimensions of anxiety and depression
Hospital Anxiety and Depression (HAD) Scale | At 1 year
  It comprises 14 items, allowing the obtaining of 2 scores out of 21 points, corresponding to the dimensions of anxiety and depression
The Short Form (36) Health Survey | Day 0
  This is a standardized test for measuring the quality of life. It includes 36 items divided into 8 dimensions (physical functioning, role limitations related to physical health, physical pain, general health, vitality [energy / fatigue], functioning or social well-being, role limitations related to mental health, Mental Health).
The Short Form (36) Health Survey | At 1,5 months
  This is a standardized test for measuring the quality of life. It includes 36 items divided into 8 dimensions (physical functioning, role limitations related to physical health, physical pain, general health, vitality [energy / fatigue], functioning or social well-being, role limitations related to mental health, Mental Health).
The Short Form (36) Health Survey | At 3 months
  This is a standardized test for measuring the quality of life. It includes 36 items divided into 8 dimensions (physical functioning, role limitations related to physical health, physical pain, general health, vitality [energy / fatigue], functioning or social well-being, role limitations related to mental health, Mental Health).
The Short Form (36) Health Survey | At 6 months
  This is a standardized test for measuring the quality of life. It includes 36 items divided into 8 dimensions (physical functioning, role limitations related to physical health, physical pain, general health, vitality [energy / fatigue], functioning or social well-being, role limitations related to mental health, Mental Health).
The Short Form (36) Health Survey | At 1 year
  This is a standardized test for measuring the quality of life. It includes 36 items divided into 8 dimensions (physical functioning, role limitations related to physical health, physical pain, general health, vitality [energy / fatigue], functioning or social well-being, role limitations related to mental health, Mental Health).
Observance of wearing the compression garment | Every week for 3 months
  Compliance with the wearing of the compression garment will be measured by the average number of hours of wearing the garment per day, which will be evaluated on the patient's statements in the experimental arm during the visits.
Tolerance of wearing the compression garment | Every week for 3 months
  The tolerance of wearing the compression garment will be assessed by recording the presence of irritation or surface skin lesion, compression felt as being too unpleasant or even unbearable by the patient in the experimental arm and leading to stopping wearing.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Detaille, Doctor, Principal Investigator — CMRRF de Kerpape
Locations (1):
- CMRRF de Kerpape, Ploemeur, Brittany Region, France

IPD SHARING:
Plan to Share IPD: No